CLINICAL TRIAL: NCT06588387
Title: Observational Retrospective Study to Assess the Use of Siponimod (Mayzent) on Patients With Secondary Progressive Multiple Sclerosis in Clinical Practice in Spain - RESYZE Study
Brief Title: A Real-world Study to Assess the Use of Siponimod in Spain to Treat Patients With Secondary Progressive Multiple Sclerosis
Acronym: RESYZE
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CBAF312AES06
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Siponimod Cohort: Patients who received at least one dose of siponimod during the drug initiation period (April 2021 to September 2022).

SUMMARY:
RESYZE was a non-interventional/observational, retrospective, multi-center study conducted in 28 public and private hospitals in Spain, assessing secondary progressive multiple sclerosis (SPMS) patients in a real-world setting. Patients underwent clinical assessments and received their standard routine medical care, as determined by their treating physicians. The study used secondary data i.e., electronic medical records (EMR) from hospitals. Patients who met the eligibility criteria were selected from the EMR of each of the sites, to include adult SPMS diagnosed patients who received at least one dose of siponimod during the start of treatment period between April 2021 and 01 September 2022, with a 12-month observation period, regardless of whether or not they continued the treatment. The study compiled data that was available in the hospital EMR from each patient up to 24 months before the first siponimod dose, and 12 months after the first siponimod dose. Data were collected for each patient at regular intervals of 6/12 months and within a window period of ±45 days, as available.

ELIGIBILITY:
Inclusion criteria:

* Patients with SPMS, as diagnosed by a physician, who started siponimod treatment at least 12 months before (during the start of the treatment period: from April 2021 to September 2022), regardless of whether they continued treatment or they did not.
* Patients who received at least 1 dose of siponimod treatment for SPMS with a 12-month observation period.
* Availability of the data for at least 12 months after siponimod initiation.

Exclusion criteria:

* Patients with any contraindication to siponimod, according to applicable Summary of Product Characteristics (SmPC).
* Patients included in any clinical trial at any moment of the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Number of Patients by Education Status | Baseline
  Education status included:
  * No studies
  * Primary education
  * Secondary education
  * Superior education
  * Unknown or missing
Number of Patients by Working Status | Baseline
  Working status included:
  * Full-time
  * Part-time
  * Retired
  * Incapacity for work
  * Medical leave
  * Unemployed
  * Student
  * Unknown or missing
Body Mass Index (BMI) | Baseline
Number of Patients by Smoking Habit | Baseline
  Smoking habits included:
  * Non-smoker
  * Smoker
  * Ex-smoker
  * Unknown or missing
Number of Patients by Alcohol Consumption | Baseline
  Alcohol consumption categories included:
  * High risk consumer
  * Low risk consumer
  * Teetotaler
  * Unknown or missing
Number of Patients by Cytochrome P450 Family 2 Subfamily C Member 9 (CYP2C9) Genotype | Baseline
  Genotype variants included:
  * CYP2C9*1*1
  * CYP2C9*1*2
  * CYP2C9*1*3
  * CYP2C9*2*2
  * CYP2C9*2*3
  * Other
Time Since Multiple Sclerosis (MS) Diagnosis | Baseline
Time Since Secondary Progressive Multiple Sclerosis (SPMS) Diagnosis | Baseline
Number of Patients by Number of Relapses in the 12 Months Before Starting Siponimod Treatment | Baseline
Number of Patients by Number of Relapses in the 24 Months Before Starting Siponimod Treatment | Baseline
Number of Patients by Number of Gadolinium T1 (Gd-T1) Lesions 24 Months Before Starting Siponimod Treatment | Baseline
Baseline Expanded Disability Status Scale (EDSS) Score at the Start of Siponimod Treatment | Baseline
  The EDSS uses an ordinal scale to assess neurologic impairment in MS based on a neurological examination. Scores in each of 7 functional systems (Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, and Cerebral) and an ambulation score were combined to determine the EDSS score. The scale ranges from 0 to 10, with 0 being normal neurological exam and 10 being death due to MS.
Number of Patients With Cognitive Decline Diagnosis | Baseline
EDSS Cognitive Subscale Score in Patients With Cognitive Decline | Baseline
  The EDSS cognitive subscale is used to grade the decrease in mentation inside the Cerebral Functional System of the EDSS scale. The scale ranges from 0 to 5, with 0 being normal (no decrease in mentation) and 5 being dementia, confusion and/or complete disorientation.
Number of Patients by Comorbidity | Baseline

SECONDARY OUTCOMES:
Number of Patients who Discontinued Siponimod Treatment | Up to 12 months
Number of Patients by Type of Siponimod Treatment Discontinuation | Up to 12 months
  Treatment discontinuation categories included temporal and permanent discontinuation.
Number of Patients by Reason for Temporal Discontinuation of Siponimod Treatment | Up to 12 months
Number of Patients by Reason for Permanent Discontinuation of Siponimod Treatment | Up to 12 months
Number of Patients Who Started a New Disease Modifying Treatment After Permanent Discontinuation of Siponimod Treatment | Up to 12 months
Number of Patients by New Disease Modifying Treatment After Permanent Discontinuation of Siponimod Treatment | Up to 12 months
Number of Patients Who Received Concomitant Treatment for Symptomatic Treatment of MS | Up to 12 months
Number of Patients by Type of Concomitant Treatment Received for Symptomatic Treatment of MS | Up to 12 months
Number of Patients by Maintenance Siponimod Dose | Up to 12 months
  Maintenance siponimod doses included 1 milligram (mg) and 2 mg.
Number of Patients who Needed a Siponimod Dose Modification | Up to 12 months
Number of Patients by Reason for Siponimod Dose Modification | Up to 12 months
Number of Patients who Needed First Dose Observation | Day 1 of the 12-month observation period
Number of Patients who Reported an Adverse Event During First Dose Observation | Day 1 of the 12-month observation period
Number of Patients who Reported an Adverse Event During Treatment With Siponimod | Up to 12 months
Number of Patients who Reported an Adverse Event of Special Interest During Treatment With Siponimod | Up to 12 months
  Adverse events of special interest included:
  * Lymphopenia
  * Macular edema
  * Bradyarrhythmia
  * Atrioventricular blockage
  * Hypertension
  * Hepatic enzymes elevation
  * Epileptic crisis
  * Infections
  * Cutaneous neoplasia
  * COVID-19
  * Death
  * Other
Number of Patients who Reported a Serious Adverse Event During Treatment With Siponimod | Up to 12 months
Number of Patients With Adverse Events Which Led to Permanent Discontinuation of Siponimod Treatment | Up to 12 months
Number of Patients With Adverse Events Which Led to Temporary Discontinuation or Dose Adjustment of Siponimod Treatment | Up to 12 months
Number of Patients With Serious Adverse Events Which Led to Permanent Discontinuation of Siponimod Treatment | Up to 12 months
Number of Patients With Serious Adverse Events Which Led to Temporary Discontinuation or Dose Adjustment of Siponimod Treatment | Up to 12 months
Number of Patients Who Died During Treatment With Siponimod | Up to 12 Months
Number of Patients by Lymphopenia Grade During Treatment With Siponimod | Baseline, Month 6, Month 12
  Lymphopenia grades:
  * Grade 1: less than lower limit of normal to 800 cells per cubic millimeters (cells/mm^3)
  * Grade 2: less than 800 to 500 cells/mm^3
  * Grade 3: less than 500 to 200 cells/mm^3
  * Grade 4: less than 200 cells/mm^3
Number of Patients With Confirmed Disability Progression During Treatment With Siponimod | Up to 12 months
  Confirmed Disability Progression was determined by an increase of at least 1 point in the Expanded Disability Status (EDSS) score if the baseline EDSS was 5.5 or less, or an increase of 0.5 points in the EDSS score if the baseline EDSS score was greater than 5.5 confirmed in a second visit performed at least 3 months apart.
  The EDSS uses an ordinal scale to assess neurologic impairment in MS based on a neurological examination. Scores in each of 7 functional systems (Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, and Cerebral) and an ambulation score were combined to determine the EDSS scores, ranging from 0 (normal) to 10 (death due to MS).
Time to First Relapse | Up to 12 months
Number of Patients Free From Relapses During the 12 Months of Treatment With Siponimod | 12 months
Number of Patients With Radiologically Detected MS Disease Activity During Treatment With Siponimod | Up to 12 months
Number of Patients With New Gd-T1 Lesions Detected After Treatment With Siponimod | Up to 12 months
Number of Patients With New or Enhanced T2 Lesions Detected After Treatment With Siponimod | Up to 12 months
Number of Patients With COVID-19 During the Study | Up to 12 months
Number of Patients by COVID-19 Vaccination Status at the Moment of COVID-19 Infection | Up to 12 months
  Vaccination status included vaccinated and not vaccinated.
Number of Patients who Required Hospitalization due to COVID-19 Infection During the Study | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States